CLINICAL TRIAL: NCT05214235
Title: A Clinical Study on the Effect of Hypoglycemic Drugs on the Prognosis of Spinal Surgery in Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, FengYafei, Associate professor, Xijing Hospital
Other Study IDs: KY20212189-C-1
Record Dates: First submitted 2021-12-30; First posted 2022-01-28 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus; Spinal Diseases
Keywords: Elective spinal surgery; Metformin; Sitagliptin; Prognosis
MeSH Terms: conditions — Diabetes Mellitus; Spinal Diseases | interventions — Hypoglycemic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Metformin: Patients who use metformin to control blood sugar level.
  Interventions: Drug: Hypoglycemic Drugs
- Sitagliptin: Patients who use sitagliptin to control blood sugar level.
  Interventions: Drug: Hypoglycemic Drugs

INTERVENTIONS:
Drug: Hypoglycemic Drugs — Patients were divided into metformin group and sitagliptin group according to the type of hypoglycemic drugs they took.

SUMMARY:
Diabetes mellitus is a group of metabolic diseases caused by multiple etiologies and characterized by chronic hyperglycemia. It seriously harms human health and has become a global public health challenge. Diabetes mellitus is present in 5% to 25% of patients undergoing spine surgery, and the prevalence has been increasing over the past decade. It is worth noting that spinal surgery for patients with diabetes has significant risks, mainly manifested in the significant increase of postoperative complications such as wound infection, delayed healing and wound hematoma, which seriously affect the long-term prognosis of patients' quality of life, spinal function and stability of internal fixation. Research shows that hypoglycemic drugs can not only control blood glucose level, but also affect the stability of nerve, bone and internal fixation, which is expected to improve the prognosis of spinal surgery in patients with diabetes. Metformin and sitagliptin are widely used hypoglycemic drugs. Studies have shown that metformin can increase bone mineral density in patients and have a protective effect on bones. Sitagliptin induces macrophage polarization of the M2 phenotype and reduces the impaired behavior of osteoblasts on titanium (TI) implants in a dose-dependent manner, thereby enhancing the bone regeneration required for successful orthopedic and dental implants in diabetic patients. However, the effects of these two drugs on the long-term prognosis of diabetic patients after spinal surgery, such as quality of life, spinal function and stability of internal fixation, have not been reported.

This investigation is a prospectie cohort study. The purpose of this study is to determine whether metformin and sitagliptin are associated with patient-reported outcomes and internal fixation stability at one year following elective spine surgery. Providers may use this information to help patients who need elective spinal surgery choose hypoglycemic drugs and to counsel patients with diabetes on expectations following spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective spinal surgery;
* Clinical diagnosis of diabetes (using the diagnostic criteria proposed by the WHO Expert Committee on Diabetes in 1999);
* Use metformin or sitagliptin;
* The age ranges from 18 to 90;
* Sign informed consent.

Exclusion Criteria:

* Acute traumatic injury;
* Patients with cerebral hemorrhage, cerebral infarction, Parkinson's disease, spinal cord transverse syndrome, spinal cord hemiere syndrome, Guillan-Barre syndrome and other neurological diseases affecting patients' somatosensory and motor;
* Combined with rheumatoid arthritis, ankylosing spondylitis and other rheumatoid arthritis;
* Patients with long-term use of glucocorticoids;
* complicated with malignant tumor;
* Pregnant women;
* Suffering from schizophrenia, bipolar disorder, hysteria and other mental diseases;
* The use of two or more than two mechanisms of hypoglycemic drugs;
* Do not sign informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A population of diabetic patients requiring elective spinal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-02-07 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Preoperative Quality of Life Score | before surgery
  Preoperative quality of life score will be performed using a Short Form-36 Health Survey (SF-36). SF-36 is a concise health questionnaire. It is widely used to measure the quality of life in the general population, evaluate the efficacy of clinical trials, and evaluate health policy. As a concise health questionnaire, SF-36 comprehensively summarized the quality of life of the respondents from nine aspects: physiological function, physical function, physical pain, general health, energy, social function, emotional function, mental health and health transition.
Quality of Life Score at 3 Months after Surgery | at 3 months after surgery
  Quality of life score at 3 months after surgery will be performed using a Short Form-36 Health Survey (SF-36). SF-36 is a concise health questionnaire. It is widely used to measure the quality of life in the general population, evaluate the efficacy of clinical trials, and evaluate health policy. As a concise health questionnaire, SF-36 comprehensively summarized the quality of life of the respondents from nine aspects: physiological function, physical function, physical pain, general health, energy, social function, emotional function, mental health and health transition.
Quality of Life Score at 6 Months after Surgery | at 6 months after surgery
  Quality of life score at 6 months after surgery will be performed using a Short Form-36 Health Survey (SF-36). SF-36 is a concise health questionnaire. It is widely used to measure the quality of life in the general population, evaluate the efficacy of clinical trials, and evaluate health policy. As a concise health questionnaire, SF-36 comprehensively summarized the quality of life of the respondents from nine aspects: physiological function, physical function, physical pain, general health, energy, social function, emotional function, mental health and health transition.
Quality of Life Score at 1 Year after Surgery | at 1 year after surgery.
  Quality of life score at 1 year after surgery will be performed using a Short Form-36 Health Survey (SF-36). SF-36 is a concise health questionnaire. It is widely used to measure the quality of life in the general population, evaluate the efficacy of clinical trials, and evaluate health policy. As a concise health questionnaire, SF-36 comprehensively summarized the quality of life of the respondents from nine aspects: physiological function, physical function, physical pain, general health, energy, social function, emotional function, mental health and health transition.
Preoperative Oswestry Disability Index (ODI) or Neck Disability Index (NDI) | before surgery
  The ODI and NDI are disease-specific questionnaires designed to gauge disability from the low back (ODI) or neck (NDI) and are scored on a 0-to-100-point scale. Values of >40 points indicate severe disability.
Oswestry Disability Index (ODI) or Neck Disability Index (NDI) at 3 Months after Surgery | at 3 months after surgery
  The ODI and NDI are disease-specific questionnaires designed to gauge disability from the low back (ODI) or neck (NDI) and are scored on a 0-to-100-point scale. Values of >40 points indicate severe disability.
Oswestry Disability Index (ODI) or Neck Disability Index (NDI) at 6 Months after Surgery | at 6 months after surgery
  The ODI and NDI are disease-specific questionnaires designed to gauge disability from the low back (ODI) or neck (NDI) and are scored on a 0-to-100-point scale. Values of >40 points indicate severe disability.
Oswestry Disability Index (ODI) or Neck Disability Index (NDI) at 1 Year after Surgery | at 1 year after surgery
  The ODI and NDI are disease-specific questionnaires designed to gauge disability from the low back (ODI) or neck (NDI) and are scored on a 0-to-100-point scale. Values of >40 points indicate severe disability.
Preoperative Visual Analogue Scale (VAS) | before surgery
  The VAS is used to assess pain. The basic method is to use a swimming scale about 10cm long, with one side marked with 10 scales, both ends of which are "0" and "10" respectively. 0 indicates no pain, and 10 indicates the most severe pain that is unbearable.
Visual Analogue Scale (VAS) at 3 Months after Surgery | at 3 months after surgery
  The VAS is used to assess pain. The basic method is to use a swimming scale about 10cm long, with one side marked with 10 scales, both ends of which are "0" and "10" respectively. 0 indicates no pain, and 10 indicates the most severe pain that is unbearable.
Visual Analogue Scale (VAS) at 6 Months after Surgery | at 6 months after surgery
  The VAS is used to assess pain. The basic method is to use a swimming scale about 10cm long, with one side marked with 10 scales, both ends of which are "0" and "10" respectively. 0 indicates no pain, and 10 indicates the most severe pain that is unbearable.
Visual Analogue Scale (VAS) at 1 Year after Surgery | at 1 year after surgery
  The VAS is used to assess pain. The basic method is to use a swimming scale about 10cm long, with one side marked with 10 scales, both ends of which are "0" and "10" respectively. 0 indicates no pain, and 10 indicates the most severe pain that is unbearable.

SECONDARY OUTCOMES:
Number of Participants with Spinal Fixation Loosening at 3 Months after Surgery | at 3 months after surgery
  Spinal fixation loosening is evaluated by anteroposterior and lateral X-ray. The evaluation criteria were: a gap of more than 1mm around the screw is considered as spinal fixation loosening.
Number of Participants with Spinal Fixation Loosening at 6 Months after Surgery | at 6 months after surgery
  Spinal fixation loosening is evaluated by anteroposterior and lateral X-ray. The evaluation criteria were: a gap of more than 1mm around the screw is considered as spinal fixation loosening.
Number of Participants with Spinal Fixation Loosening at 1 year after Surgery | at 1 year after surgery
  Spinal fixation loosening is evaluated by CT scan. The evaluation criteria were: a gap of more than 1mm around the screw is considered as spinal fixation loosening.
Number of Participants with Spinal Fusion at 3 Months after Surgery | at 3 months after surgery
  Dynamic X-ray is used to evaluate the spinal fusion. The criteria of spinal fusion:(1) there is continuous bone trabeculae passing between vertebrae with increased density; (2) The translation on the X-ray dynamic position film is less than 3mm, and the angular motion is less than 5°; (3) The bone connected to the vertebral body is constantly growing; (4) The relative displacement between adjacent spinous processes of fusion segment measured by X-ray dynamic position film is less than or equal to 2 mm.
Number of Participants with Spinal Fusion at 6 Months after Surgery | at 6 months after surgery
  Dynamic X-ray is used to evaluate the spinal fusion. The criteria of spinal fusion:(1) there is continuous bone trabeculae passing between vertebrae with increased density; (2) The translation on the X-ray dynamic position film is less than 3mm, and the angular motion is less than 5°; (3) The bone connected to the vertebral body is constantly growing; (4) The relative displacement between adjacent spinous processes of fusion segment measured by X-ray dynamic position film is less than or equal to 2 mm.
Number of Participants with Spinal Fusion at 1 Year after Surgery | at 1 year after surgery
  Dynamic X-ray is used to evaluate the spinal fusion. The criteria of spinal fusion:(1) there is continuous bone trabeculae passing between vertebrae with increased density; (2) The translation on the X-ray dynamic position film is less than 3mm, and the angular motion is less than 5°; (3) The bone connected to the vertebral body is constantly growing; (4) The relative displacement between adjacent spinous processes of fusion segment measured by X-ray dynamic position film is less than or equal to 2 mm.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Air Force Medical University (Xijing Hospital), Xi'an, Shaanxi, China